CLINICAL TRIAL: NCT03417765
Title: Double-blind, Placebo Controlled, Ascending Dose, Randomized Phase 1B/2A Study, Investigating Safety, Tolerability, PK/PD of FE 203799 in Lymphoma Patients, Undergoing Myeloablative Chemotherapy Before Autologous Transplantation
Brief Title: Safety, Tolerability, PK/PD of FE 203799 in Adults With Lymphomas
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: GlyPharma Therapeutics (Industry)
Collaborators: VectivBio AG (Industry)
Responsible Party: Sponsor
Organization: VectivBio AG (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GLY-211-2017
Record Dates: First submitted 2017-11-13; First posted 2018-01-31 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2018-10

CONDITIONS: Lymphoma, Non-Hodgkin's, Adult; Lymphoma, Hodgkin's, Adult
Keywords: gastrointestinal mucositis; myeloablative chemotherapy; autologous transplantation
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Mucositis | interventions — apraglutide

STUDY DESIGN:
Intervention Model Description: Placebo-control, ascending dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A: 5 mg (FE 203799/Placebo) (Experimental): Drug: FE 203799 Drug: BEAM Procedure: myeloablative chemotherapy Procedure: autologous stem cell transplantation
  Interventions: Drug: FE 203799
- Cohort B: 10 mg (FE 203799/Placebo) (Experimental): Drug: FE 203799 Drug: BEAM Procedure: myeloablative chemotherapy Procedure: autologous stem cell transplantation
  Interventions: Drug: FE 203799
- Cohort C: 25 mg (FE 203799/Placebo) (Experimental): Drug: FE 203799 Drug: BEAM Procedure: myeloablative chemotherapy Procedure: autologous stem cell transplantation
  Interventions: Drug: FE 203799

INTERVENTIONS:
Drug: FE 203799 — GLP-2 analogue, once weekly, subcutaneous administration

SUMMARY:
RATIONALE:

The integrity of the intestinal mucosa is a key factor for the preservation of a normal gut function. Damage of the epithelium (i.e. by chemotherapy) results in significant cellular and molecular alterations that ultimately lead to intestinal dysfunction/failure. This intestinal dysfunction manifests as several pathological processes, such as inability to absorb nutrients, intestinal inflammation, immune system dysregulation, and disequilibrium of normal intestinal microbiota leading to increased risk of infection due to bacterial translocation and septicaemia. Gastrointestinal (GI) mucositis is a well-known, frequent and debilitating side effect of most anticancer regimens with a very high incidence in hemato-oncology. The most common symptoms are nausea, vomiting, weight loss, abdominal cramps and pain, diarrhea, and electrolyte imbalance. Patients may also experience ulceration/bleeding and injury of the lining of the entire gastrointestinal tract from the esophagus to the colon. Currently no therapy is available for the prevention or treatment of GI intestinal injury. Treatment of related symptoms is limited to supportive measures to decrease diarrhea and to preventive antibiotic therapy. The GLP-2 analogue, FE 203799, has a favorable pharmacology profile for clinical development in the intended therapeutic indication of myeloablative chemotherapy-induced GI damage. The data collected from animal studies has shown that FE 203799 stimulates the proliferation of the intestinal epithelium and protects the GI mucosa from chemotherapy-induced injury. Hence, the primary pharmacologic activity of FE 203799 would promote a healthy GI microenvironment, thus preventing intestinal dysfunction and related complications.

PURPOSE: Prevention by FE 203799 of chemotherapy-induced intestinal damage and related complications in patients with lymphoma receiving Melphalan based (BEAM) myeloablative conditioning regimen followed by hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
OUTLINE:

Multi-center, double-blind, placebo-controlled, ascending dose, randomized Phase IB/2A study to assess the safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) profile of s.c. FE 203799 in patients diagnosed with Hodgkin's lymphoma (HL) or non-Hodgkin's lymphoma (NHL) undergoing Melphalan-based myeloablative chemotherapy (BEAM) followed by autologous human stem cell transplantation (AHSCT). In addition, the impact of FE 203799 on post-transplantation outcomes will be assessed. These outcomes include assessment of intestinal mucosal injury and inflammation, incidence of infection and bacteremia, development of neutropenic fever, assessment of nutritional parameters, modification of the composition of the gut microbiome, recovery of the hematopoietic system and quality of life. More specifically:

- PRIMARY OBJECTIVE: Safety and tolerability of s.c. FE 203799

- SECONDARY OBJECTIVES:

1. Determine the PK profile and dose-effect of s.c. FE 203799.
2. Determine the PD profile of s.c. FE 203799, based on the plasma concentration of citrulline (indicative of intestinal mass) and of C-Reactive Protein (CRP) (indicative of inflammation).
3. Determine the dose/response (PK/PD) relationship of s.c. FE 203799.
4. Determine the impact of treatment with s.c. FE 203799 on the incidence and severity of chemotherapy induced intestinal toxicity, as assessed by both symptomatic and visual manifestations of mucosal injury and associated complications.
5. Assess the effect of s.c. FE 203799 on the prevention of development of neutropenic fever and bacteremia.

METHODOLOGY - STUDY DESIGN The patient population will consist of adult female and male Hodgkin's or non-Hodgkin's lymphomas patients who are eligible to receive BEAM as conditioning regimen followed by autologous type AHSCT using peripheral blood or bone marrow stem cells. At the time of enrollment, patients must be in complete or partial remission following their most recent anti-neoplastic therapy. Patients are required to have available a cryopreserved autologous stem cell graft with a minimum CD34+ cell dose of 2 x 106 cells/kg.

Three ascending dose levels of FE 203799 will be investigated (5 mg, 10 mg and 25 mg), with 16 patients required per dose cohort. Patients in each dose cohort will be randomized to FE 203799 vs. Placebo in a 3:1 ratio (12 patients per dose level receiving FE 203799, and 4 patients receiving Placebo), in a double-blind manner. Randomization will occur during the screening period upon confirmation that the patient has met all inclusion and exclusion criteria. A total of 48 subjects, completing the study, is targeted for enrollment. The study will be conducted in approximately 10 clinical centers.

Eligibility will be determined at the Screening Visit following signature of the informed consent form (ICF). The inclusion and exclusion criteria will be used to qualify the patient for study entry. Within each cohort, patients will receive 4 doses of the Study Drug (FE 203799 or Placebo). As such, patients will be required to be dosed with the Study Drug the day prior the initiation of the BEAM regimen and subsequently on a weekly basis for 3 consecutive weeks after initiation of chemotherapy. Assessments performed prior to the first dose, will be considered as Baseline. Serial blood samples for determination of the plasma concentration of FE 20799/Placebo, as well as the plasma levels of citrulline and C-Reactive protein (CRP) will be obtained at pre-specified time points. During the Study, patients will be hospitalized during the duration of the conditioning chemotherapy to approximately 3 or 4 weeks post-transplantation depending on their recovery and physical condition.

All patients who received at least one treatment, will be required to return to the hospital for the End of Study Visit (Day 30 ±5 post-transplantation) and for two additional follow-up safety visits on Days 45 (±5) and 100 (±5) post-transplantation.

A Data Monitoring Committee (DMC) will convene at pre-determined timepoints, or as needed. The grading of adverse events (AEs) will be based on the Common Terminology Criteria for Adverse Events version 4.03 (CTCAE v4.03) (Grade 1 to 5).

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and non-pregnant or lactating female patients diagnosed with Hodgkin's lymphoma (HL) or non- Hodgkin's lymphoma (NHL; T- or B-cell variants) based on histological or cytological evidence.
2. Patients are eligible to receive myeloablative chemotherapy as per center eligibility criteria, followed by AHSCT.
3. Patients between 18 years and 65 years of age with a Hematopoietic Cell Transplant- Co-morbidity Index (HCT-CI) ≤5. Patients between 65 years and 70 years will be eligible if their HCT-CI score is ≤3.
4. Patients, or their legal representatives, must have the ability to read, understand and provide written informed consent prior to the initiation of any study related procedures.
5. Patients must have chemo-sensitive disease and be in partial or complete remission following the most recent anti-neoplastic therapy regimen, according to the Lugano revision of the International Working Group (IWG) response criteria [1].
6. Patients must have available a cryopreserved autologous hematopoietic stem cell graft containing ≥ 2.0 x 106 cryopreserved CD34+ cells/kg.
7. Patients must have a Karnofsky score ≥ 70%.
8. Patients must have adequate hepatic function as evidenced by bilirubin ≤ upper limit of normal (ULN), unless felt to be related to Gilbert's syndrome or hemolysis; patients must also have AST and ALT ≤ 1.5 x ULN and alkaline phosphatase ≤ 2.5 x ULN.
9. Patients must have an estimated or measured creatinine clearance ≥ 30 ml/min/1.73 m2 by the Cockcroft-Gault equation.
10. Patients must have left ventricular ejection fraction ≥ 50%.
11. Patients must have forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1) and diffusing capacity corrected for hemoglobin (DLCOc) ≥ 50% of predicted.
12. Patients must have recovered from the effects of any prior chemotherapy, radiotherapy or surgery; for patients who have been on monoclonal antibody therapy, at least one half-life or 4 weeks (whichever is longer) should have elapsed prior to the first scheduled day of dosing with FE 203799.
13. A female recipient of childbearing potential must meet the following criteria:

    1. Participant has a negative pregnancy test at Screening.
    2. Participant agrees to use one of the accepted contraceptive regimens from at least 14 days prior to the first administration of the Study Drug, during the study and for at least 90 days after the last dose of the Study Drug. An acceptable method of contraception includes one of the following:

       * Abstinence from heterosexual intercourse
       * Systemic contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
       * Intrauterine device (with or without hormones)
       * Diaphragm with spermicidal gel
       * Condom with spermicide gel
14. A male patient, with sexual partners who are pregnant, possibly pregnant, or who could become pregnant, agrees to use one of the accepted contraceptive regimens throughout the entire duration of the study and until at least 3 months after the last drug administration. An acceptable method of contraception includes one of the following:

    * Abstinence from heterosexual intercourse
    * Condom with spermicide

Exclusion Criteria:

1. Patient is unable or unwilling to give informed consent.
2. Patients who are unable to comply with the treatment protocol including appropriate supportive care, follow-up and tests.
3. Patients with known hypersensitivity to FE 203799, or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions to any drugs.
4. Patients with an active infection or with a fever ≥38.5oC within 3 days of the first scheduled day of dosing.
5. Patients who had an autologous stem cell transplant within 24 months.
6. Patients who had an available cryopreserved autologous graft with a CD34+ cell count of < 2 x 106/kg.
7. Patients undergoing AHSCT for conditions other than lymphoma.
8. Presence of a malignancy other than the one for which the transplant is being performed (except for baso-cellular skin carcinoma).
9. Patients who are receiving investigational therapies or who have been treated with investigational therapies or investigational devices within 30 days prior to the first scheduled day of dosing with FE 203799.
10. Patients with cardiovascular congestive heart failure, unstable angina pectoris, cardiac arrhythmias requiring a pacemaker; myocardial infarction within the past six months; stroke within the past 6 months; or uncontrolled hypertension.
11. Patients with mean QTcF values of >450 msec (in males) or >470 msec (in females) following ECGs conducted in triplicate 5 minutes apart from each other; patients who are known to have congenital prolonged QT syndromes, including patients who are already on medication known to cause prolonged QT intervals on ECG.
12. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 220 msec, QRS < 60 msec, QRS >119 msec) on the screening ECG or other clinically significant ECG abnormalities.
13. Patients with history or presence of GI tract cancer, polyps, ulcerative colitis, Crohn's disease, coeliac disease, tropical sprue, etc.
14. Presence of active pancreatic disease.
15. Presence of active liver disease (i.e. cirrhosis; bilirubin > ULN; transaminases > 1.5 x ULN; alkaline phosphatase > 2.5 x ULN).
16. Presence of autoimmune disease.
17. Patients with suicidal tendency or clinically relevant psychiatric diseases or substance abuse.
18. Positive results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HbsAG (B) (hepatitis B)) or anti-Hepatitis C Virus (HCV (C)) tests.
19. Any abnormal condition or laboratory result that is considered by the PI capable of altering patient's condition or study outcome.
20. Patients who are pregnant or lactating.
21. Patients who are unwilling to use appropriate contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Day -8 to Day 100
  Adverse events as assessed by CTCAE v4.03

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of FE 203799 | Day -8 to Day 13
  Cmax in ng/ml
Cumulative area under the plasma concentration (AUC) time curve from 0-168 hours of FE 203799 | Day -8 to Day 13
  AUC0-168 in ng*hr/ml
Cumulative area under the plasma concentration (AUC) from time zero to infinity of FE 203799 | Day -8 to Day 13
  AUC0-inf in ng*hr/ml
Terminal elimination half-life (T1/2) of FE 203799 | Day -8 to Day 13
  T1/2 in hours
Apparent total body clearance (CL) of the drug from plasma of FE 203799 | Day -8 to Day 13
  CL in ml/hr
Apparent volume of distribution (Vz) of FE 203799 during terminal phase | Day -8 to Day 13
  Vz in ml
Biomarker assessment for gut healing | Day -8 to Day -1, Day 1 to Day 14 and Day 30
  Plasma concentration of citrulline (ng/ml)
Biomarker assessment for gut inflammation | Day -8 to Day -1, Day 1 to Day 14 and Day 30
  Plasma concentration of C-Reactive Protein (ng/ml)
Assessment of infection - Incidence and duration of fever | Day -8 to Day 20 and Day 30
  Body temperature ≥38.2oC
Assessment of infection - Incidence and duration of neutropenic fever | Day -8 to Day 20 and Day 30
  Development of fever when absolute neutrophil count (ANC) ≤ 0.5 x 109 and body temperature ≥ 38.2 ◦C for two consecutive values over a 30 minute period of time; or ANC < 0.5 x 109 and body temperature ≥ 38.5◦C at any single timepoint
Incidence of microbiologically detected infection | Day 5 to Day 15
  Blood cultures once daily
Assessment of gastrointestinal mucositis and related clinical symptoms | Day -8 to Day 20 and Day 30
  Grading as by the CTCAE v4.03
Assessment of gastrointestinal mucositis by video-capsule endoscopy | Day -8, Day 6 and Day 20
  Gastrointestinal damage assessed by the Lewis Score; this is evaluation of villous edema, ulcers and stenosis graded collectively; Normal < 135, Mild 135-790, Moderate - severe ≥790
Assessment of nutrients absorption | Days -8, -1, 6, 13 and 30
  Body weight (kg)
Assessment of nutrients absorption | Days -8, 0, 3, 6, 9, 12, 15, 18
  Assessment of duration of parenteral nutrition (L)
Assessment of nutrients absorption | Days -8, 0, 3, 6, 9, 12, 15, 18
  Assessment of caloric intake (calories)
Microbiome composition | Once a week over 4 weeks
  Determination of microbial populations by genomic analysis (relative abundance of taxonomic levels)
Time to neutrophil and platelet engraftment | Day-8 and then on Days -2, 5, 12 and 30
  Hematological analysis
Assessment of quality of life | Days -8, -1, 6, 13 and 30
  Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Masior, Study Director — VectivBio AG

IPD SHARING:
Plan to Share IPD: No